CLINICAL TRIAL: NCT03284294
Title: The Influence of Vitamin D Supplementation on Serum Brain Derived Neurotrophic Factor Level and Cognitive Function in Schizophrenia Treated With Atypical Antipsychotic
Brief Title: Influence of Vitamin D Supplementation on Serum BDNF Level and Cognitive Function in Schizophrenia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Principal Investigator, Tuti Kurnianingsih, Principal Investigator, Universitas Padjadjaran
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PS-201709.01
Record Dates: First submitted 2017-09-04; First posted 2017-09-15 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Oral placebo daily for 8 weeks
  Interventions: Drug: Placebo
- Vitamin D (Active Comparator): Vitamin D Cholecalciferol 2000 IU oral daily for 8 weeks
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — cholecalciferol 2000 IU oral daily for 8 weeks
  Arms: Vitamin D
Drug: Placebo — Oral placebo daily for 8 weeks
  Arms: Placebo

SUMMARY:
The objective of the study is to evaluate the influence of vitamin D supplementation on Serum Brain Derived Neurotrophic Factor level and cognitive function in schizophrenia treated with atypical antipsychotic. Methods: The investigator will use randomized controlled trial design. 40 chronic schizophrenia patients with vitamin D insufficiency or deficiency treated with atypical antipsychotic, will be randomly assign (1:1 ratio) to receive either daily oral cholecalciferol 2000 IU or placebo for 8 weeks. Assessment of BDNF serum and cognitive function will be performed at baseline and after 8 weeks period.

ELIGIBILITY:
Inclusion Criteria:

* Chronic schizophrenia
* Serum 25(OH)D level below 30 ng/ml
* Deficit in cognitive functions

Exclusion Criteria:

* Hypercalcemia
* Hepatic or renal failure
* Obese
* Metabolic syndrome

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-04-15 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function | At the end of week 8
  cognitive function as measured with standard cognitive battery

SECONDARY OUTCOMES:
BDNF serum level | At the end of week 8
  BDNF serum level as measured with ELISA method

IPD SHARING:
Plan to Share IPD: No